CLINICAL TRIAL: NCT02573376
Title: Antiviral Pharmacology and Adherence in Drug Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Denver Health and Hospital Authority (Other); National Institute on Drug Abuse (NIDA) (NIH); Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 15-0809; 1R01DA040499-01 (NIH)
Record Dates: First submitted 2015-06-03; First posted 2015-10-09 (Estimated); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: HEPATITIS C; Virus, Human Immunodeficiency
Keywords: HIV; Hepatitis C; Drug Abuse; Hepatitis C Virus; sofosbuvir; ledipasvir; pharmacology; pharmacokinetics
MeSH Terms: conditions — Hepatitis C; Acquired Immunodeficiency Syndrome; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sofosbuvir/Ledipasvir with Directly Observed Therapy (DOT) (Other): Participants randomized to vDOT will be provided a smart phone with cellular service and will be pre-programmed with the mobile phone-based video application and contact information for study personnel.
  Interventions: Behavioral: Directly Observed Therapy
- Sofosbuvir/Ledipasvir with Wirelessly Observed Therapy (WOT) (Other): Participants on WOT will be provided the Wisepill portable medication dispenser.
  Interventions: Behavioral: Wirelessly Observed Therapy

INTERVENTIONS:
Behavioral: Directly Observed Therapy
  Other Names: DOT
  Arms: Sofosbuvir/Ledipasvir with Directly Observed Therapy (DOT)
Behavioral: Wirelessly Observed Therapy
  Other Names: WOT
  Arms: Sofosbuvir/Ledipasvir with Wirelessly Observed Therapy (WOT)

SUMMARY:
Approximately one half of all Americans living with Hepatitis C virus (HCV) are drug users, yet they are the least likely to receive HCV treatment. Drug users are presumed non-adherent and therefore denied potentially life-saving therapy. This assumption can only be confirmed or dispelled through prospective pharmacologic and adherence studies in this population. Such studies would be greatly enhanced by an objective, quantitative measure of adherence which does not currently exist in the HCV field. Through the work proposed in this application, sixty HIV/HCV co-infected drug users will be treated with direct acting antiviral agents (DAA) and randomized to receive directly observed DAA therapy (DOT) vs. no directly observed therapy (no-DOT). Patients randomized to no-DOT will have wirelessly observed therapy (WOT) which involves use of a portable medication dispenser that sends a signal to a server with the date and time when the dispenser is opened. In Aim 1, DAA concentrations will be compared in those randomized to DOT vs. no-DOT. DAA pharmacokinetics will also be defined accounting for clinical factors like degree of hepatic impairment and use of concomitant recreational and antiretroviral drugs. The goal is to quantify adherence in this population and the effect of variable adherence on drug concentrations. In Aim 2, DAA concentrations (plasma, cellular, hair) will be linked with adherence patterns identified using WOT and DOT. The goal is to identify a drug concentration biomarker that predicts adherence in this population. In Aim 3, the relationship between DAA adherence (as measured by WOT and DOT and drug concentrations) and rate of cure will be established. The goal is to define the degree of adherence needed for HCV cure.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* HIV-infected men and women
* Chronic HCV infection as documented by quantifiable HCV RNA
* HCV genotype 1, 4, 5, 6
* 18-70 years of age
* Willingness and ability to comply with study procedures, including DOT, WOT, and biweekly clinic visits
* Considered an active drug user by HCV provider and self-reported drug use within the past month

Exclusion Criteria:

* Glomerular filtration rate < 30 mL/min/1.73 m2
* Receipt of prior HCV treatment and radiographic, histologic, or clinical evidence of cirrhosis
* Decompensated liver disease (i.e., ascites, history of esophageal variceal bleeding, hepatic encephalopathy)
* Medications not recommended per the SOF/LDV prescribing information (e.g., tipranavir and other P-gp inducers, tenofovir disoproxil fumarate plus cobicistat, rosuvastatin, amiodarone)
* Any medical condition that in the opinion of the investigators will make it challenging to adhere to the study protocol, such as unstable heart disease or cancer
* Chronic Hepatitis B virus Infection
* For females, active pregnancy or any intent to become pregnant
* For both sexes, an unwillingness to use contraception during the study period
* On parole or impending sentencing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Compare each individual's modeled estimate of ledipasvir and metabolites of sofosbuvir (GS-331007 and GS-331007-TP) steady state concentrations (Css) from non-linear mixed effects modeling to Css in subjects receiving DOT vs. WOT. | 12 weeks
Quantify GS-331007-TP concentrations in dried blood spots as a function of adherence (doses taken/doses prescribed). | 12 weeks
Estimate the probability of HCV cure as a function of adherence using logistic regression. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer J Kiser, PharmD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States